CLINICAL TRIAL: NCT03754881
Title: Efficacy of 8-week Supervision in Home Based Pulmonary Rehabilitation
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sei Won Lee, Associate Professor, Asan Medical Center
Other Study IDs: 2018-0964
Record Dates: First submitted 2018-11-21; First posted 2018-11-27 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Pulmonary rehabilitation — In this study, we'll educate pulmonary rehabilitation to patients and make reservation for re-visiting outpatients clinics with PR diary after 8 weeks.
  we want to confirm whether patients, who perform home based PR during more than 30 minutes in 3 days per week, present improved dyspnea score or quality of life compared with non-compliance group.

SUMMARY:
In korea, it is not easy to practice standard pulmonary rehabilitation (PR). in this study, we'll educate PR to patients and make reservation for re-visiting outpatients clinics with PR diary. we want to confirm whether patients, who perform home based PR during more than 30 minutes in 3 days per week, present improved dyspnea score or quality of life compared with non-compliance group.

ELIGIBILITY:
Inclusion Criteria:

* forced expiratory volume-one second / forced vital capacity < 0.7 in post-bronchodilator pulmonary function test
* adults 40 years or older
* no history of acute exacerbation within 4 weeks
* no history of education for pulmonary rehabilitation within 6 months
* no change of medication for chronic obstructive pulmonary disease within 4 weeks
* dyspnea more than Modified Medical Research Council grade 0

Exclusion Criteria:

* adults under 40 years old
* no consent
* history of acute exacerbation within 4 weeks
* history of education for pulmonary rehabilitation within 6 months
* change of medication for chronic obstructive pulmonary disease within 4 weeks
* dyspnea only Modified Medical Research Council grade 0
* comorbidity, including cardiovascular disease, orthopedic disease, neurologic disease, optic disease, uncontrolled hypertension
* enrolled other clinical trial
* on long term oxygen therapy

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic obsturctive pulmonary disease in Asan Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-05-05 (Actual); Study Completion 2020-09-06 (Actual)

PRIMARY OUTCOMES:
Change from basline Chronic obstructive pulmonary disease (COPD) assessment Test (CAT) at 8 weeks | 8 weeks
  Self reported Patient-completed questionnaire assessing globally the impact of COPD (cough, sputum, dyspnea, chest tightness) on health status. Each item is scored 0-5, yielding a total between 0 and 40

SECONDARY OUTCOMES:
change from 6 minutes walk test at 8 weeks | 8 weeks
  This test measures the distance that a patient can quickly walk on a flat, hard surface in a period of 6 minutes (the 6MWD).
Change from the Short Form 36 Health survey (SF-36), version 2.0 at 8 weeks | 8 weeks
  a 36-item, patient-reported survey of patient health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability.
Change from BODE index at 8 weeks | 8 weeks
  BODE index include forced expiratory volume-one second, 6 minutes walk distance, modified Medical Research Council dyspnea scale, body mass index. The BODE Index is used to predict mortality.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pulmonary and Critical Care Medicine and Clinical Research Center for Chronic Obstructive Airway Diseases, Asan Medical Center, University of Ulsan College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lee JH, Lee HY, Jang Y, Lee JS, Oh YM, Lee SD, Lee SW. Efficacy of Unsupervised Home-Based Pulmonary Rehabilitation for Patients with Chronic Obstructive Pulmonary Disease. Int J Chron Obstruct Pulmon Dis. 2020 Sep 28;15:2297-2305. doi: 10.2147/COPD.S268683. eCollection 2020. PMID 33061347